CLINICAL TRIAL: NCT04092712
Title: A Phase 1, Open-label Study to Assess the Absorption, Metabolism, Excretion, and Mass Balance of Oral [14C]-CTP-543 in Healthy Adult Male Subjects
Brief Title: Study Evaluating Pharmacokinetics and Mass Balance of [14C]-CTP-543 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP543.1004
Record Dates: First submitted 2019-09-05; First posted 2019-09-17 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Mass Balance; Radiolabeled; Pharmacokinetics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Product (Experimental): [14C]-CTP-543
  Interventions: Drug: [14C]-CTP-543

INTERVENTIONS:
Drug: [14C]-CTP-543 — Single dose of radiolabeled CTP-543 (approximately 75 μCi) administered as an oral solution

SUMMARY:
This study will assess the absorption, metabolism, excretion, mass balance, safety, and tolerability of a single oral administration of [14C]-CTP-543 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 55 years, inclusive (healthy is determined by medical evaluation, including medical history, full physical examination, vital signs, electrocardiogram, and clinical laboratory tests)
* Body Mass Index of 18.0 to 32.0 kg/m2
* Continuous non smoker who has not used nicotine containing products for at least 3 months prior to dosing and throughout the study

Exclusion Criteria:

* Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening
* Infection with hepatitis B or hepatitis C viruses
* History of irregular bowel movements
* History of herpes zoster
* A positive tuberculosis test at screening or history of incompletely treated or untreated tuberculosis
* History or presence of alcoholism or drug abuse within the past 2 years prior to dosing
* Participation in another clinical study within 30 days prior to dosing

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Mass balance: Calculation of percent of total radioactivity recovered in urine | From time zero up to 96 hours post-dose following oral administration of [14C]-CTP-543 up to Day 15
Mass balance: Calculation of percent of total radioactivity recovered in feces | From time zero up to 96 hours post-dose following oral administration of [14C]-CTP-543 up to Day 15
CTP-543 PK: Cmax | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Maximum plasma concentration
CTP-543 PK: Tmax | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Time for Cmax
CTP-543 PK: t1/2 | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
CTP-543 PK: AUClast | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration (Clast)
CTP-543 PK: AUCinf | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to infinity
CTP-543 PK: CL/F | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes).
CTP-543 PK: Vz/F | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Apparent volume of distribution following oral administration
CTP-543 metabolite PK: Cmax | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Maximum plasma concentration
CTP-543 metabolite PK: Tmax | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Time for Cmax
CTP-543 metabolite PK: t1/2 | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
CTP-543 metabolite PK: AUC0-last | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to time of the last quantifiable concentration (Clast)
CTP-543 metabolite PK: AUCinf | Pre-dose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Area under the plasma concentration time profile from time 0 to infinity
Total [14C]: urine | Pre-dose up to 336 hours post-dose
  Total radioactivity excreted into the urine from time zero to the time of last measurable concentration following oral administration of [14C]-CTP-543
Total [14C]: feces | Pre-dose up to 336 hours post-dose
  Total radioactivity excreted into the feces from time zero to the time of last measurable concentration following oral administration of [14C]-CTP-543
Total radioactivity in whole blood | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose
Total radioactivity in plasma | Pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-dose

SECONDARY OUTCOMES:
Adverse events | Screening up to Day 15
  Number of adverse events, which are any untoward medical occurrence regardless of attribution to study drug in a participant who received study drug
Number of Participants With Clinically Significant Change From Baseline in Heart Rate | Screening, Pre-dose, 2, 8, 48 hours post-dose
  Heart rate measured in beats per minute (bpm)
Number of Participants With Clinically Significant Change From Baseline in Blood Pressure | Screening, Pre-dose, 2, 8, 48 hours post-dose
  Blood pressure measured in millimeters of mercury (mmHg)
Number of Participants With Clinically Significant Change From Baseline in Respiratory Rate | Screening, Pre-dose, 2, 8, 48 hours post-dose
  Respiratory rate measured in breaths per minute
Number of Participants With Clinically Significant Change From Baseline in Temperature | Screening, Pre-dose, 2, 8, 48 hours post-dose
  Temperature measured in Celsius (°C)
Number of Participants With Clinically Significant Change From Baseline in Hematology | Screening, Check-in, 8, 24 hours postdose
Number of Participants With Clinically Significant Change From Baseline in Serum Chemistry | Screening, Check-in, 8, 24 hours postdose
Number of Participants With Clinically Significant Change From Baseline in Coagulation | Screening, Check-in, 8, 24 hours postdose
Number of Participants With Clinically Significant Change From Baseline in Urinalysis | Screening, Check-in, 8, 24 hours postdose
Number of Participants With Clinically Significant Changes to the Physical Examination | Screening up to Day 15
  Clinically significant changes to the physical examination
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram - P Wave | Screening, Pre-dose, 48 hours post-dose
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram - QRS Complex | Screening, Pre-dose, 48 hours post-dose
Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram - QT Interval | Screening, Pre-dose, 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States